CLINICAL TRIAL: NCT02521779
Title: Dietary Fat Affects Postprandial Serum Endotoxin Concentration in Healthy Adults
Brief Title: The Role of Dietary Fat on Postprandial Endotoxemia in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, James Hollis, Associate Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14-020; 2014-67017-21778 (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2015-07-28; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Endotoxemia
Keywords: Inflammation; Endotoxemia; Lipopolysaccharide; Diet; Fat; Postprandial
MeSH Terms: conditions — Endotoxemia; Inflammation; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test Meal Saturated Fat (Experimental): Saturated-fat Treatment Meal
  Interventions: Other: Saturated-fat Treatment Meal
- Test Meal N-6 Fat (Experimental): N-6 fat Treatment Meal.
  Interventions: Other: N-6 fat Treatment Meal
- Test Meal N-3 Fat (Experimental): N-3 fat Treatment Meal.
  Interventions: Other: N-3 fat Treatment Meal
- Test Meal Low-fat (Experimental): Low-fat Treatment Meal.
  Interventions: Other: Low-fat Treatment Meal

INTERVENTIONS:
Other: Low-fat Treatment Meal — Isocaloric test meal that provided 20% fat.
  Arms: Test Meal Low-fat
Other: Saturated-fat Treatment Meal — Isocaloric test meal that provided 35% fat with saturated fat (16 g).
  Arms: Test Meal Saturated Fat
Other: N-3 fat Treatment Meal — Isocaloric test meal that provided 35% fat with n-3 (DHA = 500mg)
  Arms: Test Meal N-3 Fat
Other: N-6 fat Treatment Meal — Isocaloric test meal that provided 35% fat with n-6 (7.4 g).
  Arms: Test Meal N-6 Fat

SUMMARY:
The purpose of this study was to determine the effect of different dietary fats (saturated or unsaturated) on postprandial endotoxemia and systemic low grade acute inflammation. The investigators hypothesized that meals rich in saturated or n-6 fatty acids would increase postprandial endotoxemia but meals high in n-3 fatty acids would decrease postprandial endotoxemia.Participants were recruited via email and randomized to treatment meal in this single-blind, cross-over study. Each test session participants reported to the laboratory right away in the morning. An indwelling catheter was inserted into the participant non-dominant arm by a qualified nurse and a baseline blood draw was taken. The participant was then provided with one of four test meals (a porridge-type meal containing a different dietary fat), which they ate in entirety within 15 minutes. The participants remained in the laboratory for the next five and a half hours and were not allowed to consume any food or drink except water. During this time, further blood draws were taken at intervals of one hour for a total of five hours after the consumption of the test meal. Collected blood was processed on-site and the serum fraction collected and tested for endotoxin, inflammatory biomarkers, and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years old;
* Willingness to eat test meals;
* Body mass index ≥ 19.9 ±0.8 and ≤ 24.9 ±0.8;
* Weight stable (< 2 kilogram weight change in the previous 3 months)

Exclusion Criteria:

* Presence of acute or chronic disease;
* Use of tobacco products;
* Consumes more than 21 units of alcohol per week;
* Use of anti-inflammatory medication;
* History suggestive of macronutrient malabsorption

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Serum endotoxin concentration | Change from baseline every one hour, up to five hours

SECONDARY OUTCOMES:
Serum concentration of biomarkers of inflammation | Change from baseline every one hour, up to five hours
Serum concentration of triglycerides, glucose, and non-esterified fatty acids | Change from baseline every one hour, up to five hours

CONTACTS AND LOCATIONS:
Overall Officials: James H Hollis, PhD, Principal Investigator — Iowa State University
Locations (1):
- Nutrition and Wellness Research Center, Ames, Iowa, United States

REFERENCES:
- [Background] Erridge C, Attina T, Spickett CM, Webb DJ. A high-fat meal induces low-grade endotoxemia: evidence of a novel mechanism of postprandial inflammation. Am J Clin Nutr. 2007 Nov;86(5):1286-92. doi: 10.1093/ajcn/86.5.1286. PMID 17991637
- [Background] Fritsche KL. The science of fatty acids and inflammation. Adv Nutr. 2015 May 15;6(3):293S-301S. doi: 10.3945/an.114.006940. Print 2015 May. PMID 25979502
- [Background] Mani V, Hollis JH, Gabler NK. Dietary oil composition differentially modulates intestinal endotoxin transport and postprandial endotoxemia. Nutr Metab (Lond). 2013 Jan 10;10(1):6. doi: 10.1186/1743-7075-10-6. PMID 23305038
- [Derived] Lyte JM, Gabler NK, Hollis JH. Postprandial serum endotoxin in healthy humans is modulated by dietary fat in a randomized, controlled, cross-over study. Lipids Health Dis. 2016 Nov 5;15(1):186. doi: 10.1186/s12944-016-0357-6. PMID 27816052